CLINICAL TRIAL: NCT04439383
Title: Risk Stratification for Hospital-Acquired Venous Thromboembolism in Medical Patients: a Prospective Cohort Study
Brief Title: Risk Stratification for Venous Thromboembolism in Hospitalized Medical Patients
Acronym: RISE
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); University Hospital, Geneva (Other); University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: RISE
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Venous Thromboembolism; Venous Thromboses; Pulmonary Embolism; Deep Vein Thrombosis; Embolism and Thrombosis; Mobility Limitation; Hospital Acquired Condition
Keywords: Venous thromboembolism; Pulmonary embolism; Deep vein thrombosis; Risk factor; Hospital-acquired; Mobility; Accelerometry
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Embolism and Thrombosis; Mobility Limitation; Iatrogenic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hospital-acquired venous thromboembolism (HA-VTE) is one of the leading preventable causes of in-hospital mortality, but prevention of VTE in hospitalized medical patients remains challenging, as preventive measures such as pharmacological thromboprophylaxis (TPX) need to be tailored to individual thrombotic risk.

The broad objective of this project is to improve VTE prevention strategies in hospitalized medical patients by prospectively examining VTE risk factors (including mobility) and comparing existing risk assessment models.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Admitted for hospitalization >24 hours on a general internal medicine ward
* Informed consent as documented by signature

Exclusion Criteria:

* Need for therapeutic anticoagulation (e.g., atrial fibrillation)
* Life expectancy <30 days
* Insufficient proficiency of the German or French language
* Unwilling to provide informed consent
* Prior enrolment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely ill adult patients hospitalized for at least 24h in general internal medicine of the participating tertiary care hospitals
Sampling Method: Probability Sample
Enrollment: 1353 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism | Within 90 days of initial hospital admission
  Symptomatic, objectively confirmed fatal and non-fatal hospital-acquired venous thromboembolism, including symptomatic distal and proximal deep vein thrombosis and pulmonary embolism after hospital admission

SECONDARY OUTCOMES:
Venous thromboembolism | During the initial hospitalization, an average of 7 days
  Symptomatic, objectively confirmed fatal and non-fatal hospital-acquired venous thromboembolism, including symptomatic distal and proximal deep vein thrombosis and pulmonary embolism during hospitalization
All-cause mortality | During hospitalization (an average of 7 days) and up to 90 days of initial hospital admission
  All-cause mortality (all causes of death will be considered)
Major bleeding | During hospitalization (an average of 7 days) and up to 90 days of initial hospital admission
  Major bleeding will be defined as fatal bleeding, symptomatic bleeding at critical sites (intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, pericardial, or intramuscular with compartment syndrome), or bleeding with a reduction of hemoglobin of at least 20 g/L or bleeding leading to transfusion of 2 or more units of packed red blood cells according to the definition of the International Society on Thrombosis and Haemostasis
Clinically relevant non-major bleeding | During hospitalization (an average of 7 days) and up to 90 days of initial hospital admission
  Clinically relevant non-major bleeding, defined as overt bleeding that does not meet criteria for major bleeding but is associated with a medical intervention, unscheduled physician contact (visit or telephone call), or pain or impairment of activities of daily life
Patient autonomy in the activities of daily living | At discharge (an average of 7 days after initial hospital admission) and at 90 days after admission
  Patient autonomy in the activities of daily living as assessed by the modified Barthel Index
Length of hospital stay | within 90 days of initial hospital admission
  Length of hospital stay, defined as the time/date of discharge minus time/date of admission at the hospital ward
Subsequent hospitalizations | Within 90 days of initial hospital admission
  Subsequent hospitalization, defined as hospital readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Christine Baumgartner, MD, MAS, Principal Investigator — Inselspital, Bern University Hospital; Marie Méan, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois, University Hospital of Lausanne
Locations (3):
- Switzerland (3):
  - Inselspital, Bern University Hospital, Bern
  - Geneva University Hospital, Geneva
  - University Hospital of Lausanne, Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choffat D, Farhoumand PD, Jaccard E, de la Harpe R, Kraege V, Benmachiche M, Gerber C, Leuzinger S, Podmore C, Truong MK, Dumans-Louis C, Marti C, Reny JL, Aujesky D, Rakovic D, Limacher A, Rossel JB, Baumgartner C, Mean M. Risk stratification for hospital-acquired venous thromboembolism in medical patients (RISE): Protocol for a prospective cohort study. PLoS One. 2022 May 24;17(5):e0268833. doi: 10.1371/journal.pone.0268833. eCollection 2022. PMID 35609087